CLINICAL TRIAL: NCT05911997
Title: Comparison of MTC01 vs FMT for the Treatment of Recurrent Clostridioides Difficile Infection
Brief Title: MTC Versus FMT in for RCDI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ari M Grinspan, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-23-00563; 1R01DK130337-01A1 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Clostridiodies Difficile Infections
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Four different interventions
Masking Description: All open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Dose MTC 01 (Experimental): High dose MTC 01 is 10 x 11 CFU slurry to be administered via colonoscopy
  Interventions: Drug: MTC 01
- Low Dose MTC 01 (Experimental): Low Dose MTC 01 is 10 x 10 CFU slurry to be administered via colonoscopy
  Interventions: Drug: MTC 01
- Low dose Fecal Microbiota Transplantation (FMT) (Active Comparator): High dose FMT is 10 x 11 CFU slurry to be administered via colonoscopy
  Interventions: Drug: Fecal Microbiota Transplantation (FMT)
- High Dose Fecal Microbiota Transplantation (FMT) (Experimental): Low dose FMT is 10 x 10 CFU slurry to be administered via colonoscopy
  Interventions: Drug: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Drug: MTC 01 — Slurry to be administered via colonoscopy
  Arms: High Dose MTC 01; Low Dose MTC 01
Drug: Fecal Microbiota Transplantation (FMT) — Stool from a healthy donor is blended with salt water and made into a liquid solution rich in bacteria. This solution is sprayed into the recipient's colon during a colonoscopy
  Other Names: Full spectrum FMT from a single donor
  Arms: High Dose Fecal Microbiota Transplantation (FMT); Low dose Fecal Microbiota Transplantation (FMT)

SUMMARY:
Investigating four different treatment of MTC or FMT

DETAILED DESCRIPTION:
The purpose of this research study is to compare two different treatments for patients with recurrent Clostridiodies difficile infections: MTC01 vs fecal microbiota transplantation (FMT). FMT is the transfer of bacteria from a healthy donor's colon to a recipient's colon. To do this, stool from a healthy donor is blended with salt water and made into a liquid solution rich in bacteria. This solution is sprayed into the recipient's colon during a colonoscopy. This treatment is now considered standard medical care for recurrent Clostridioides difficile infections.

One FMT dose contains the entire collection of microbes in a healthy donor and is made up of billions of microbes. Each dose of FMT is different from the next and it is unknown exactly what microbes are present in each dose.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18 years and older
* Able and willing to provide written informed consent
* History of recurrent CDI defined as 2 episodes of CDI occurring within the previous 6 months (inclusive of the current episode)
* Subjects with a qualifying recurrent CDI episode, defined as:

  * History of diarrhea (>=3 unformed stools per day for 2 or more consecutive days that is clinically consistent with CDI
  * Documented positive stool test by local laboratory for toxigenic C. difficile (toxin EIA or PCR-based testing) for the current CDI episode within 60 days prior to randomization.
  * Received a course of standard-of-care (SOC) CDI antibiotics for the most recent CDI episode (for 10 to 42 days, with exact duration, antibiotic type and dose at the discretion of the Investigator)
  * Demonstrated adequate clinical response, defined as <= 3 unformed stools per day for 2 or more consecutive days during SOC CDI antibiotics prior to randomization.
* CDI symptoms started within 60 days prior to randomization.

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding or are planning to become pregnant during the study.
* Women with reproductive potential should use a reliable method of birth control:

  * Consistent use of an approved hormonal contraception (birth control pill/patches, rings); An intrauterine device (IUD); Contraceptive injection (Depo-Provera); Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam); Sexual abstinence (no sexual intercourse) or Sterilization
* Known or suspected toxic megacolon, ileus or bowel obstruction at the time of enrollment.
* Subjects with active gastroenteritis due to infectious causes other than CDI
* Subjects with allergies to ingredients present in the investigational product
* Prior participation in studies of investigational live biotherapeutic products or FMT within the last 6 months.
* Major gastrointestinal surgery within the last 3 months before enrollment.
* Use of drugs that alter gut motility.
* History of acute leukemia or hematopoietic stem cell transplantation or myelosuppressive chemotherapy within 2 months prior to enrollment.
* Unable or unwilling to undergo a colonoscopy
* Inpatient status, though patients can be screened while inpatients, the must be outpatient for the planned colonoscopy.
* Anticipated immediate or upcoming surgery within 30 days
* Need for continued non-anti-CDI antibiotic therapy
* History of total proctocolectomy
* Patients who are unable to give informed consent
* Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
* Severe food allergy (anaphylaxis or anaphylactoid-like reaction)
* Life expectancy < 6 months
* Unable to adhere to protocol requirements
* Patient who have received an FMT in the past year
* Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines that it will put the subject at greater risk from FMT
* Clinically significant abnormal lab values including but not limited to WBC >15 x 103/mm3, ANC <0.5 x 103/mm3, or laboratory evidence of acute kidney injury at Investigator's discretion, at screening
* If a patient is heavily immunosuppressed and is negative for CMV or EBV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-related serious adverse events (SAE) as assessed by NIH grading | up to 24 weeks
  Number of serious adverse events per NIH grading indications. Grade 1-5, where grade 3-5 are considered severe.
  1. Mild
  2. Moderate
  3. Severe
  4. Life threatening
  5. Death Serious Adverse Event (SAE):
  Any adverse event that:
  * Results in death
  * Is life threatening, or places the participant at immediate risk of death from the event as it occurred
  * Requires or prolongs hospitalization
  * Causes persistent or significant disability or incapacity
  * Results in congenital anomalies or birth defects
  * Is another condition which investigators judge to represent significant hazards
Number of participants with treatment-related adverse events as assessed by CTCAE 5.0 | up to 24 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0, grade 1-2, where higher grades indicate higher levels of impairment.
  1. Mild
  2. Moderate
  3. Severe
  4. Life threatening
  5. Death

SECONDARY OUTCOMES:
Percent of patients who develop Clostridioides difficile (C difficile) | within 8 weeks
  Recurrence of Clostridioides difficile (C difficile) within 8 weeks of receiving treatment. The stool C difficile toxin test detects harmful substances produced by the C difficile bacterium . This infection is a common cause of diarrhea after antibiotic use. Abnormal results mean that toxins produced by C difficile are seen in the stool and are causing diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Grinspan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will not be shared with patients. However aggregate data will be shared with the NIH and for publications. The DSMB is within mount Sinai.